CLINICAL TRIAL: NCT01732939
Title: Phase II Study of Neoadjuvant Chemotherapy Regimen Choice in Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Affiliated to Military Medical Science, Beijing (Other)
Responsible Party: Sponsor
Other Study IDs: 307BCNeo-01
Record Dates: First submitted 2012-10-10; First posted 2012-11-26 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- AT: Docetaxel 75 mg/m2, day 1 or paclitaxel 175mg/m2 day 1 plus Epirubicin 75 mg/m2, day 1 or doxorubicine 50mg/m2 day 1 for 6-8 cycles
- AT-NP: docetaxel 75mg/m2,day 1 or paclitaxel 175mg/m2,day 1 plus doxorubicine 50mg/m2,day 1 or epirubicin 75mg/m2, day 1,for3-4 cycles then switch to vinorelbine 25mg/m2, day 1 and day 8 plus cisplatinum 75mg/m2, day 1 for 3-4 cycles

SUMMARY:
The study purpose is to observe which neoadjuvant chemotherapy regimens is the better for invasive breast cancer. The neoadjuvant chemotherapy regimen is sustained anthracyclines plus taxanes or from anthracyclines plus taxanes to vinorelbine plus cisplatinum.

DETAILED DESCRIPTION:
The investigators hope to get preliminary results for the breast cancer patients who are given different neoadjuvant chemothetapy regimens. The patients are randomized two chemotherapy regimens. One is anthracyclines plus taxanes for 6-8 cycles,the other is anthracyclines plus taxanes for 3-4 cycles ,then switch tovinorelbine plus cisplatinum for 3-4 cycles.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of invasive ductal or lobular breast cancer.
* Previously untreated (no chemotherapy or hormonal therapy or radiation therapy) invasive breast cancer.
* no anti-Her2 therapy if HER2 positive ( defined as 3+ IHC or FISH positive)
* Performance Status ECOG <2
* Age > 18 years
* Tumor > 2.0 cm by MRI and/or sonographic or clinical exam measurements.or Karnofsky >50%
* Lab test :

  * Absolute neutrophil count > 1,500/mm3

    * Total Bilirubin ≤ 2×ULN
    * AST and ALT ≤ 2.5×ULN
  * serum creatinine ≤ 1.5×ULN

Exclusion Criteria:

* Pregnant or breast feeding patients are excluded
* stage Ⅳ breast cancer
* History of non-breast malignancies within the 5 years prior to study entry, except for the following: carcinoma in situ of the cervix, carcinoma in situ of the colon,melanoma in situ, and basal cell and squamous cell carcinomas of the skin
* uncontrolled cardiac disease
* Active infection or chronic infection requiring chronic suppressive antibiotics
* History of hypersensitivity reaction to investigating drugs

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: diaganosis of invasive breast cancer, tumor size > 2.0cm by MRI or ultrasound or clinical examination.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2012-05; Primary Completion 2013-12 (Actual); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
pathological complete response rate | one year

SECONDARY OUTCOMES:
clinical response rate, safety | one year

CONTACTS AND LOCATIONS:
Overall Officials: Zefei Jiang, MD, Principal Investigator — Hospital Affiliated Military Medical Science
Locations (1):
- Hospital affiliated academy military medical science, Beijing, Beijing Municipality, China